CLINICAL TRIAL: NCT02259283
Title: Prospective Study on the Feasibility and Results of the Treatment of Idiopathic Achalasia With the POEM (Per Oral Endoscopic Myotomy) Technique
Brief Title: Prospective Study on the Feasibility and Results of POEM in Idiopathic Achalasia
Acronym: POEM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, Chief of Clinical research Project, Istituto Clinico Humanitas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POEM-ICH
Record Dates: First submitted 2014-09-29; First posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Achalasia
Keywords: achalasia; per oral endoscopic myotoymy; endoscopy
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Achalasia (Experimental): Patients (age 18-75 years old) with diagnosis of achalasia, without megaesophagus or colonic esophagus, will undergo POEM with the hybrid knife.
  Interventions: Device: Hybrid Knife

INTERVENTIONS:
Device: Hybrid Knife — POEM (Per oral endoscopic myotoymy) technique performed with the hybrid knife which combines injection and cutting in the same device.

SUMMARY:
Treatment options for achalasia include endoscopic dilations and surgical myotomy. Recently the POEM (Per oral endoscopic myotoymy) technique has been described. Patients undergo myotomy under endoscopic control. It has advantage over endoscopic dilation since myotomy is performed, and has advantage over surgery because it is performed endoscopically, thus is less invasive. One potential disadvantage in respect to surgery may be that it may determine higher rates of post-operative reflux. The purpose of this study is to prospectively assess the feasibility of PEOM in our Center with the new hybrid knife, and clinical results at 1, 3 and 12 months.

This is a prospective, phase II study. Ten patients (age 18-75 years old) with diagnosis of achalasia, without megaesophagus or colonic esophagus, will be included for the POEM procedure.

This study will last about 2 years. The aim is the feasibility, security and success rate of POEM for achalasia. Patients will be followed for at least one year.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years
* Manometric diagnosis of achalasia
* Eckardt score more than 3
* Informed consent

Exclusion Criteria:

* Increased surgical risk for important comorbidities,
* Pseudoachalasia
* Mega-esophagus (more than 7 cm) and or sigmoid esophagus,
* Previous esophageal or gastric surgery (with the exception of gastric perforation)
* Inability of completing the questionnarie
* Inability to keep a commitment for follow-up
* Esophageal diverticulum

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-12; Primary Completion 2014-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Feasibility | 24 months
  Percentage of patients with successful POEM
Clinical Success | 24 months
  A reduction of 2 or more points in the Eckardt score, that determines a score of 3 or more in 24 months.

SECONDARY OUTCOMES:
Quality of Life | 24 months
  Quality of life as measured by questionnaires (SF36 and l'EORTC QLQ-OES24) that will be administered to the patients at 3 and 12 months.
Adverse events | 24 months
  Post-operative adverse events (perforation, bleeding, infection, aspiration, etc)
Reflux disease | 24 months
  Reflux disase as diagnosed clinically (HRQL questionnarie) or by 24-hour pH-metry
Treatment failure | 24 months
  Percentages of patients in which other interventions for dysphagia are required after the first POEM.
Efficacy | 24 months
  Basal and post-treatment pressure of the lower esophageal sphincter, as measured by manometry and esophageal follow-through.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Repici, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Endoscopy Unit, Humanitas Research Hospital, Rozzano, Milano, Italy

REFERENCES:
- [Background] Eckardt VF, Aignherr C, Bernhard G. Predictors of outcome in patients with achalasia treated by pneumatic dilation. Gastroenterology. 1992 Dec;103(6):1732-8. doi: 10.1016/0016-5085(92)91428-7. PMID 1451966
- [Background] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937
- [Background] Swanstrom LL, Kurian A, Dunst CM, Sharata A, Bhayani N, Rieder E. Long-term outcomes of an endoscopic myotomy for achalasia: the POEM procedure. Ann Surg. 2012 Oct;256(4):659-67. doi: 10.1097/SLA.0b013e31826b5212. PMID 22982946